CLINICAL TRIAL: NCT00812669
Title: An Open-label Phase II Study of the Efficacy and Safety of the Combination of Fludarabine, Cyclophosphamide and Rituximab in Patients With Chronic Lymphocytic Leukaemia Who Are Newly Diagnosed, Have Relapsed or Are Resistant to First-Line Treatment
Brief Title: CLL-Irl Study. CTRIAL-IE (ICORG) 07-01, V7
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTRIAL-IE (ICORG) 07-01; CTRIAL-IE (ICORG) 07-01; 2008-001250-40; EU-20898
Record Dates: First submitted 2008-12-19; First posted 2008-12-22 (Estimated); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Leukemia
Keywords: B-cell chronic lymphocytic leukemia; refractory chronic lymphocytic leukemia; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — pegfilgrastim; Rituximab; Cyclophosphamide; fludarabine phosphate; Cytogenetic Analysis; In Situ Hybridization, Fluorescence; Gene Expression Profiling; Flow Cytometry

ARMS (1):
- Fludarabine, Cylophosphamide and Rituximab (Experimental)
  Interventions: Biological: pegfilgrastim; Biological: rituximab; Drug: cyclophosphamide; Drug: fludarabine phosphate; Genetic: cytogenetic analysis; Genetic: fluorescence in situ hybridization; Genetic: gene expression analysis; Genetic: mutation analysis; Genetic: protein expression analysis; Other: flow cytometry; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: pegfilgrastim
Biological: rituximab
Drug: cyclophosphamide
Drug: fludarabine phosphate
Genetic: cytogenetic analysis
Genetic: fluorescence in situ hybridization
Genetic: gene expression analysis
Genetic: mutation analysis
Genetic: protein expression analysis
Other: flow cytometry
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fludarabine and cyclophosphamide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Giving fludarabine together with cyclophosphamide and rituximab may kill more cancer cells.

PURPOSE: This phase II trial is studying giving fludarabine together with cyclophosphamide and rituximab to see how well it works in treating patients with chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the efficacy, in terms of complete remission rate, of fludarabine phosphate, cyclophosphamide, and rituximab in patients with chronic lymphocytic leukemia.

Secondary

* Determine the time to treatment failure (TTF) in these patients.
* Determine the overall survival of these patients until 10th January 2019.
* Assess the predictive value of immunophenotype, hypermutation analysis, and FISH in determining TTF and OS in these patients.
* Determine the safety profile of this regimen.

OUTLINE: This is a multicenter study.

Patients receive fludarabine IV over 30 minutes or orally and cyclophosphamide IV or orally on days 1-3 and pegfilgrastim subcutaneously on day 4. Starting on course 2, patients receive rituximab IV on day 1. Treatment repeats every 28 days for up to 6* courses in the absence of disease progression or unacceptable toxicity.

NOTE: *Patients achieving negative minimal residual disease receive 4 courses of treatment.

Blood samples are collected periodically for biomarker analysis. Samples are analyzed for protein expression (i.e., CD38, CD20, and ZAP70) by flow cytometry; quantitative immunoglobulins, β2-microglobulin, and T-cell subsets by electrophoresis; IgVH mutation status; and cytogenetics (i.e., +12, del 13q, del 11q, and del 17p) by FISH.

After completion of study therapy, patients are followed every 6 months for 5 years and then annually until 10th January 2019.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of chronic lymphocytic leukemia

  * Stage I-IV disease (Binet stage progressive A, B, C)
  * CD5 and CD23 positive
  * Untreated OR relapsed/resistant disease after combination chemotherapy or rituximab
  * No 17p deletion

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Life expectancy > 1 year
* Creatinine clearance ≥ 50 mL/min
* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other concurrent malignancy except for noninvasive cervical cancer or localized nonmelanomatous skin cancer
* No history of anaphylaxis to mouse-derived humanized monoclonal antibody
* No other severe concurrent (e.g., cardiac or pulmonary) diseases or mental disorders that could interfere with ability to participate in the study

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 0 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Actual)
Dates: Start 2008-08-18 (Actual); Primary Completion 2019-11-21 (Actual); Study Completion 2019-11-21 (Actual)

PRIMARY OUTCOMES:
Complete remission rate by NCI response criteria and minimal residual disease (MRD) analysis | A formal assessment of response by NCI Criteria (Appendix 3) with the addition of assessment of minimal residual disease in the marrow and if relevant assessment of bulky disease by CT scanning will be made after 4 +/-6 courses of therapy.

SECONDARY OUTCOMES:
Time to treatment failure (TFF) | A clinical assessment of response will be made after 4 courses of therapy, Patients with evidence of progressive disease will stop therapy and will be deemed to have failed treatment.
Overall survival | Until 10th January 2019
Predictive value of immunophenotype, FISH, and hypermutation analysis in determining TTF and OS | See description
  Timing and type of response assessment
  During chemotherapy. A clinical assessment of response will be made after 4 courses of therapy. Patients with evidence of progressive disease will stop therapy and will be deemed to have failed treatment. A formal assessment of response by NCI Criteria (Appendix 3) with the addition of assessment of minimal residual disease in the marrow and if relevant assessment of bulky disease by CT scanning will be made after 4 +/-6 courses of therapy.
  Following chemotherapy. Disease assessment after the end of therapy will involve a history(recording B-symptoms), complete physical examination, full blood count and blood MRD analysis every 6 months for 5 years and then annually until 10th of January 2019 or until disease progression.
Acute and chronic toxicity as assessed by NCI criteria | A formal assessment of response by NCI Criteria (Appendix 3) with the addition of assessment of minimal residual disease in the marrow and if relevant assessment of bulky disease by CT scanning will be made after 4 +/-6 courses of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Vandenberghe, MD, Principal Investigator — St. James's Hospital, Ireland
Locations (7):
- Ireland (7):
  - Tallaght University Hospital, Dublin, Leinster
  - Cork University Hospital, Cork, Munster
  - St. James's Hospital, Dublin
  - University College Hospital, Galway
  - University Hospital Limerick, Limerick
  - Midland Regional Hospital at Tullamore, Tullamore
  - Waterford Regional Hospital, Waterford

REFERENCES:
- [Derived] Appleby N, O'Brien D, Quinn FM, Smyth L, Kelly J, Parker I, Scott K, Cahill MR, Crotty G, Enright H, Hennessy B, Hodgson A, Leahy M, O'Leary H, O'Dwyer M, Hayat A, Vandenberghe EA. Risk adjusted therapy in chronic lymphocytic leukemia: a phase II cancer trials Ireland (CTRIAL-IE [ICORG 07-01]) study of fludarabine, cyclophosphamide, and rituximab therapy evaluating response adapted, abbreviated frontline therapy with FCR in non-del(17p) CLL. Leuk Lymphoma. 2018 Jun;59(6):1338-1347. doi: 10.1080/10428194.2017.1376746. Epub 2017 Sep 19. PMID 28925785
- See also: Summary of Clinical trial findings published in "Leukemia and Lymphoma". — https://www.ncbi.nlm.nih.gov/pubmed/28925785